CLINICAL TRIAL: NCT00000721
Title: An Escalating Dose Tolerance Trial of BG8962 (rCD4) in Patients Who Are HIV Antibody Positive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 066; 11040 (Registry Identifier: DAIDS ES Registry Number); 066 Extension
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Infusions, Intravenous; Injections, Intramuscular; Injections, Intravenous; Injections, Subcutaneous; Dose-Response Relationship, Drug; Drug Evaluation; Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — CD4 Antigens

INTERVENTIONS:
Drug: CD4 Antigens

SUMMARY:
To determine the maximal safe daily dose of BG8962 (rCD4) which can be administered by continuous subcutaneous infusion (CSCI) over 24 hours; to determine the pharmacokinetics of BG8962 when it is administered by intramuscular and subcutaneous routes; and to look for dose related antiviral activity determined by quantitation of infectious HIV peripheral blood leukocytes (PBLs) and plasma, and by monitoring the blood levels of viral p24 antigen (when present), CD4+ T-cells, and Beta-2- microglobulin. Recombinant soluble CD4 protein (rCD4) is a drug that has been produced by genetic engineering techniques. In laboratory studies, rCD4 binds to HIV and reduces its ability to enter the cell, thus inhibiting its reproduction. Before rCD4 can be tested for therapeutic effectiveness in HIV-infected patients, it is necessary to determine the maximum dose that can be tolerated by humans. AMENDED: To date, Biogen's original sequence recombinant soluble CD4 and Biogen's natural sequence recombinant soluble CD4 have both been referred to as recombinant soluble CD4 (rsCD4). In order to distinguish between these two products, a change in nomenclature has been made. In this protocol, whenever the original sequence CD4 molecule is referred to, it is called recombinant soluble T4 (rsT4). Whenever the natural sequence molecule (currently under study in this protocol) is referred to, it is called BG8962 or rCD4. Whenever the drug is discussed generically, it is referred to as rsCD4.

DETAILED DESCRIPTION:
Recombinant soluble CD4 protein (rCD4) is a drug that has been produced by genetic engineering techniques. In laboratory studies, rCD4 binds to HIV and reduces its ability to enter the cell, thus inhibiting its reproduction. Before rCD4 can be tested for therapeutic effectiveness in HIV-infected patients, it is necessary to determine the maximum dose that can be tolerated by humans. AMENDED: To date, Biogen's original sequence recombinant soluble CD4 and Biogen's natural sequence recombinant soluble CD4 have both been referred to as recombinant soluble CD4 (rsCD4). In order to distinguish between these two products, a change in nomenclature has been made. In this protocol, whenever the original sequence CD4 molecule is referred to, it is called recombinant soluble T4 (rsT4). Whenever the natural sequence molecule (currently under study in this protocol) is referred to, it is called BG8962 or rCD4. Whenever the drug is discussed generically, it is referred to as rsCD4.

The initial dose level is the highest dose previously established with other patients in this trial to be safe when administered intramuscularly (IM). Dose escalation is by semilogarithmic steps. A shift from IM injection to continuous subcutaneous infusion (CSCI) is necessitated by the volume of drug which is administered as part of the escalation dose. Three groups of eight patients each are treated as follows. The first group of 8 patients receives BG8962 daily and consists of two cohorts of four patients each. One cohort receives BG8962 as an IM injection. The second cohort receives BG8962 as a continuous 24 hour infusion. All patients in this group are treated for 12 weeks. The second dosing group of 8 patients receive daily BG8962 by CSCI for 12 weeks. The third group of 8 patients receive BG8962 by CSCI for 6 weeks. Every two weeks during the study the following tests and evaluations are done: Blood chemistry, hematology, urinalysis with microscopic exam, and T-cells and T-cell subsets.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Nystatin or clotrimazole for suppression of oral thrush.
* Aerosolized pentamidine for Pneumocystis prophylaxis in Group A patients.
* Trimethoprim / sulfamethoxazole for Pneumocystis prophylaxis in patients who are hematologically stable on trimethoprim / sulfamethoxazole.

Patients must have:

* Group A: AIDS and symptoms defined in disease status.
* Group B: AIDS related complex (ARC) and symptoms defined in disease status.

Exclusion Criteria

Co-existing Condition:

Patients with the following disease or conditions are excluded:

* Malignancies other than Kaposi's sarcoma.
* AIDS dementia.
* Opportunistic infections requiring ongoing therapy except oral thrush suppression with nystatin or clotrimazole or Pneumocystis prophylaxis in Group A patients.
* Significant organ system dysfunction including:
* Granulocytopenia with a granulocyte count < 1000 cells/mm3.
* Thrombocytopenia - < 75000 platelets/mm3.
* Anemia with a hemoglobin < 9.5 g/dl.
* Renal dysfunction - creatinine > 2 mg/dl.
* Hepatic dysfunction with enzymes or bilirubin > 3 x upper limit of normal.

Patients with the following are excluded:

* Preexisting antibodies to rCD4.
* Malignancies other than Kaposi's sarcoma.
* AIDS-dementia complex.
* Opportunistic infections requiring ongoing therapy.
* Significant organ system dysfunction.
* Inability to sign voluntarily the consent form.

Prior Medication:

Excluded:

* Recombinant soluble CD4 protein (rCD4).
* Excluded within 30 days of study entry:
* Immunomodulatory therapy or agent with anti-HIV activity.
* Chemotherapy.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiotherapy.

Active illicit drug use or alcohol abuse at time of entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85
Dates: Study Completion 1991-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Schooley RT, Study Chair; Merigan TC, Study Chair
Locations (1):
- Stanford CRS, Palo Alto, California, United States